CLINICAL TRIAL: NCT01456299
Title: Target-controlled Infusion of Remifentanil for Laryngeal Mask Airway Insertion During Sevoflurane Induction in Adults
Brief Title: Laryngeal Mask Airway (LMA) Insertion With Sevoflurane and Remifentanil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Jeong Kwak, Associate Professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AJIRB-MED-CT4-11-045; AJIRB-MED-CT4-11-045 (Registry Identifier: Ajou University IRB)
Record Dates: First submitted 2011-10-19; First posted 2011-10-20 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Laryngismus
Keywords: laryngeal mask airway; insertion; sevoflurane; remifentanil
MeSH Terms: conditions — Laryngismus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): The control group, which received an infusion of normal saline.
  Interventions: Drug: Control
- Remifentanil 1 (Active Comparator): "Remifentanil 1": "The R1 group, which received a target effect-site remifentanil concentration of 1 ng/ml.
  Interventions: Drug: Remifentanil 1
- Remifentanil 2 (Active Comparator): "Remifentanil 2": "The R2 group, which received a target effect-site remifentanil concentration of 2 ng/ml.
  Interventions: Drug: Remifentanil 2

INTERVENTIONS:
Drug: Remifentanil 1 — "Remifentanil 1": "The R1 group, which received a target effect-site remifentanil concentration of 1 ng/ml.
  Other Names: R1
  Arms: Remifentanil 1
Drug: Control — The control group, which received an infusion of normal saline
  Other Names: Placebo
  Arms: Control
Drug: Remifentanil 2 — "Remifentanil 2": "The R2group, which received a target effect-site remifentanil concentration of 2 ng/ml.
  Other Names: R2
  Arms: Remifentanil 2

SUMMARY:
The purpose of this study was to determine the most suitable effect-site concentration of remifentanil for the LMA insertion during inhaled induction with 8% sevoflurane in adults.

DETAILED DESCRIPTION:
For practical purposes, opioids with the ability to suppress upper airway reflexes have been used to facilitate insertion of the LMA during anaesthesia induction. To date, however, there have been no published reports addressing the use of remifentanil to facilitate LMA insertion during sevoflurane inhalation induction in adults. Therefore, the purpose of this study was to determine the most suitable effect-site concentration of remifentanil target-controlled infusion (TCI) for the LMA insertion during inhaled induction with 8% sevoflurane in adults.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients, aged 18-60 with ASA physical status I or II, who were scheduled to minor elective surgery (< 1 h) were considered for the study

Exclusion Criteria:

- Exclusion criteria were allergies to the study drugs, a history of gastric reflux, a history of drug abuse, obesity (body mass index > 30 kg/m2) and suspected difficult airway

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, MD,PhD, Study Director — Ajou University School of Medicine; Jong Yeop Kim, MD, PhD, Study Director — Ajou Universiy School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, South Korea

REFERENCES:
- [Background] Sivalingam P, Kandasamy R, Madhavan G, Dhakshinamoorthi P. Conditions for laryngeal mask insertion. A comparison of propofol versus sevoflurane with or without alfentanil. Anaesthesia. 1999 Mar;54(3):271-6. doi: 10.1046/j.1365-2044.1999.00663.x. PMID 10364865

RESULTS

PARTICIPANT FLOW:
Groups:
- Remifentanil 1: The R1 group, which received a target effect-site remifentanil concentration of 1 ng/ml
  control: Patients received a normal saline only
- Control: The control group, which received an infusion of normal saline
  remifentanil 1: The patients received an infusion of remifentanil
- Remifentanil 2: The R2 group, which received a target effect-site remifentanil concentration of 2 ng/ml
  remifentanil 2: Patients received no remifentanil
Period: Overall Study
Arm/Group | Remifentanil 1 | Control | Remifentanil 2
Started | 34 | 34 | 34
Completed | 34 | 33 | 33
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: no differences in patient characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Remifentanil 1 | Remifentanil 2 | Total
Number analyzed (Participants) | 33 | 34 | 33 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (11) | 37 (12) | 38 (11) | 38 (11)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 34 | 33 | 100
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 18 | 60
  Male | 13 | 12 | 15 | 40
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 33 | 34 | 33 | 100

OUTCOME MEASURES:

1. Primary Outcome: LMA Insertion Condition
Description: The pre-determined effect-site concentration of remifentanil or normal saline was administered according to the patient's group.LMAs were size #3 for women and #4 for men.The conditions of the LMA insertion were graded on a three point scale using six variables (mouth opening, ease of LMA insertion, swallowing, coughing and gagging, head and body movements, laryngospasm). Each of these variables was rated as excellent, intermediate or poor.
Time Frame: at that time on LMA insertion only
Measure: Number; unit: participants
Arm/Group | Control | Remifentanil 1 | Remifentanil 2
Number analyzed (Participants) | 33 | 34 | 33
participants
  Excellent | 14 | 21 | 24
  Intermediate | 7 | 5 | 3
  Poor | 12 | 8 | 6

2. Secondary Outcome: Frequency of Apnea
Description: If prolonged apnoea (> 30 s) developed, manual ventilation was assisted. And record the frequency of apnea on each group
Time Frame: baseline, 30sec after drug injection
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control | Remifentanil 1 | Remifentanil 2
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes